CLINICAL TRIAL: NCT06043323
Title: A Phase II Study of Axicabtagene Ciloleucel, an Anti-CD19 Chimeric Antigen Receptor (CAR) Tcell Therapy, in Combination With Radiotherapy (RT) in Relapsed/Refractory Follicular Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0087; NCI-2023-07173 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine phosphate; Prednisone; Diphenhydramine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Axicabtagene Ciloleuce (Experimental): Participants will first have a procedure to collect your white blood cells that will be used to make axicabtagene ciloleucel. Then participatns will receive radiation therapy, followed by conditioning chemotherapy and 1 infusion of axicabtagene ciloleucel.
  Interventions: Drug: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine phosphate; Drug: Prednisone; Drug: Diphenhydramine; Drug: Acetaminophen

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — Given by IV (vein)
Drug: Cyclophosphamide — Given by IV (vein)
  Other Names: Cytoxan®; Neosar®
Drug: Fludarabine phosphate — Given by IV (vein)
Drug: Prednisone — Given by IV (vein)
Drug: Diphenhydramine — Given by IV (vein)
  Other Names: Benadryl®
Drug: Acetaminophen — Given by IV (vein)
  Other Names: Tylenol®; Dorcol®; Feverall; Panadol; APAP; N-Acetyl-P-Aminophenol; Paracetamo; Ofirmev™

SUMMARY:
To learn about the safety of a drug called axicabtagene ciloleucel given in combination with radiation therapy to patients with relapsed/refractory FL.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of this study is to determine the safety of standard of care axicabtagene ciloleucel with bridging radiotherapy (RT) in patients with relapsed or refractory follicular lymphoma, as assessed by the incidence of grade 3 or higher cytokine release syndrome (CRS) within 30 days after chimeric antigen receptor (CAR) T-cell infusion.

Secondary Objectives:

* Establish the rates of CRS and ICANS in patients treated with CAR T-cell therapy and radiation
* Determine complete response rate (CR) at approximately 1 month post CAR T-cell ---therapy
* Determine complete response rate (CR) at approximately 6 month post CAR T-cell ---therapy
* Determine the overall response rate (ORR)
* Determine the duration of response (DOR)
* Determine progression free survival (PFS)
* Determine overall survival (OS)

Exploratory Objectives:

* Assess the impact of tumor burden as measured by metabolic tumor volume and total lesion glycolysis on PET/CT on response following CAR T-cell infusion
* Assess T-cell fitness from blood samples by flow cytometry and ssRNAseq prior to and after bridging RT
* Perform immune profiling of blood samples for T-cell subsets prior to and after bridging RT
* Assess cytokine profile after infusion

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be considered for inclusion if they meet all of the following criteria:

* Men and women 18 years of age or older
* Histologically proven FL (Grade 1-3A) on most recent biopsy, history of transformed follicular lymphoma permitted at clinician discretion)
* Patients with follicular lymphoma must have disease that has relapsed or is refractory to 2 or more prior lines of systemic therapy
* (ECOG) performance status of 0-2
* Medically appropriate for CAR-T cell therapy: adequate organ function CrCL >/= 45 mL/min/m2, hemoglobin level ≥ 8 g/dl, serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) levels ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 x ULN if documented liver involvement, baseline oxygen saturation levels (SpO2) ≥92% on room air
* Have at least 1 measurable lesion on imaging, defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) and ≥1 cm on CT, MRI, or clinical exam.
* Prior radiation therapy is permitted provided normal tissue tolerance is not exceeded
* Female of child-bearing potential (FOCBP, defined below) must have a negative pregnancy test within 1 week of simulation for RT
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of other (non B-cell lymphoma) invasive malignancy requiring active therapy (systemic therapy, radiation, or surgery) within the past 3 years, excluding non-melanomatous skin cancer
* Women of childbearing potential who are pregnant
* Women who are breastfeeding and unwilling to discontinue prior to lymphodepleting chemotherapy and for 12 months following lymphodepleting chemotherapy and CAR-T cell infusion
* Urgent need for bridging chemotherapy or rituximab between apheresis and CAR T cell product infusion (steroids permitted)
* Additional RT would exceed standard organ at risk constraints
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Uncontrolled fungal, bacterial, or viral infection requiring intravenous antimicrobials for management. Urinary tract infection and uncomplicated bacterial pharyngitis is permitted if responding to active treatment. Recent COVID19 infection is permitted if patient is deemed medically stable for CAR-T cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org